CLINICAL TRIAL: NCT03557606
Title: A Case Series Evaluating the Use of Bone Marrow Concentrate for the Treatment of Alar, Accessory, and Transverse Ligament Injuries
Brief Title: Case Series on Using Bone Marrow Concentrate for Alar Ligament Injuries
Status: Withdrawn | Type: Observational
Why Stopped: Collecting data as part of a Patient Registry; redundant study.
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RSI2017-CASE01
Record Dates: First submitted 2018-05-09; First posted 2018-06-15 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Craniocervical Injuries
Keywords: CCJ; Bone Marrow Concentrate; Stem Cell Therapy; Alar Ligament; Transverse Ligament
MeSH Terms: conditions — Trauma, Nervous System

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alar treatment with BMC: Patients with CCJ instability that receive Alar treatment with BMC using anterior approach.
  Interventions: Procedure: Alar treatment with BMC using anterior approach

INTERVENTIONS:
Procedure: Alar treatment with BMC using anterior approach — Patients with CCJ instability will undergo a bone marrow aspiration of approximately 30-60 cc. Platelet rich plasma (PRP) and platelet lysate (PL) will be derived from the bone marrow aspirate and later mixed with the bone marrow cell layer. While under TIVA anesthesia, the injectate is then injected under fluoroscopy into the area in need of treatment using an anterior approach through the posterior oropharynx with direct visualization of the injection site via endoscopy. The alar, transverse, and accessory ligaments are the target areas to be treated with the bone marrow concentrate.

SUMMARY:
A prospective case series of 200 patients who have been treated with Bone Marrow Concentrate using anterior approach through posterior oropharynx for treating alar, accessory, and transverse injuries for patients with craniocervical junction instability.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the clinical outcomes for patient who are treated with with bone marrow concentrate (BMC) using an anterior approach through the posterior oropharynx for treating alar and transverse ligament injuries as part of their clinical care. The case series will observe pre and post-treatment subject-reported clinical outcomes. Secondary objectives include evaluation of post-treatment complications, adverse events, re-injections, and surgical intervention, change in use of pain medications, and changes on post treatment imaging.

The treatment consists of patients undergoing a bone marrow aspiration of approximately 30-60 cc. Platelet rich plasma (PRP) and platelet lysate (PL) will be derived from the bone marrow aspirate and later mixed with the bone marrow cell layer. While under anesthesia, the injectate is then injected under fluoroscopy into the area in need of treatment using an anterior approach through the posterior oropharynx.

One of the challenges of treating the upper cervical ligaments through injection is that they can't be accessed from the posterior due to obstruction from the cervical spinal cord. The investigator's group has developed an injection technique using an anterior approach through the posterior oropharynx, which allows direct access to the ligaments for injection. The goal of this study is to evaluate the effectiveness of this procedure in CCJ instability patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) Voluntary signature of the IRB approved Informed Consent, 2) Skeletally mature Male or Female ages 18 to 65 3) Disabling symptoms of headache, dizziness, neck pain, or other neuro-musculoskeletal symptoms, that based on physical exam or diagnostic blocks is attributable to the upper cervical spine for >12 months 4) Symptoms exacerbated by activity and relieved by rest 5) Failed all conservative care 6) Hasn't responded long-term to:

  1. C0-C3 facet injections
  2. Upper cervical prolotherapy or PRP into the posterior stabilizing ligaments (nuchal, supraspinous, interspinous ligaments) 7) Considered a likely cervical fusion candidate 8) Imaging (one of the three)

  <!-- -->

  1. Upper cervical MRI showing decreased signal in alar, transverse, PAOM, AAOM, or Tectorial membrane
  2. DMX showing 2 mm or greater lateral overhang of C1 on C2 in lateral bending open mouth view or a V shaped ADI in flexion of increased ADI in flexion
  3. Upper cervical rotatory CT that shows excessive C0-C1 rotation 9) Exam is c/w upper cervical injury (i.e. tenderness along upper cervical facet joints and/or musculature/skull base, good anesthetic block response (>50% pain relief) to C0-C3 intra-articular facet injections, proprioceptive difficulties) 10) Is independent, ambulatory, and can comply with all post-operative evaluations and visits 11) Patient states strong desire to avoid surgery

Exclusion Criteria:

* 1) Unable to tolerate injections due to central sensitization (i.e. significant intolerance to manual therapy such as massage, activity such as physical therapy, or an exaggerated pain response to prior injection therapy)

  2) Previous neck surgery that has caused chronic neck pain or radiculopathy 3) Prior epidural or other milligram dose steroid injection in any area or other neck injection therapy within the past 6 months 4) Physical infirmity that is incompatible with the procedure and/or anesthesia required for same 5) Unable to tolerate the injection position 6) Abnormal anatomy seen on MRI imaging that would make the procedure higher risk (e.g. congenital atlanto-axial fusion, atlas assimilation, upper cervical fracture or surgical fusion)

  7) Inflammatory or auto-immune based pathology (e.g., rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout, pseudo gout) 8) Quinolone or Statin induced myopathy/tendinopathy

  9) Condition represents a worker's compensation case 10) Currently involved in a health-related litigation procedure 11) Is pregnant 12) Bleeding disorders 13) Currently taking anticoagulant or immunosuppressive medication 14) Allergy or intolerance to study medication 15) Use of and significant physical dependence on a chronic opioid (>20 mg oxycodone equivalent per day) 16) Documented history of drug abuse within six months of treatment 17) Any other condition, that in the opinion of the investigator, that would preclude the patient from enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking treatment at an orthopedic pain management and regenerative medicine clinic.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Headache Impact Test score change from baseline | Change from Baseline to 6 months
  The within patient mean change from baseline to 6 months in Headache Impact Test scores. Scale of 36-78; HIT-6 scores 36-49 (little to no impact), HIT-6 scores 50-55 (moderate impact), HIT-6 scores 56-59 (substantial impact), HIT-6 scores 60-78 (severe impact ).

SECONDARY OUTCOMES:
Headache Impact Test score change from baseline | Change from baseline to 12 months
  The within patient mean change from baseline to 6 months in Headache Impact Test scores. Scale of 36-78; HIT-6 scores 36-49 (little to no impact), HIT-6 scores 50-55 (moderate impact), HIT-6 scores 56-59 (substantial impact), HIT-6 scores 60-78 (severe impact ).
Neck Disability Index score change from baseline | Change from baseline to 6 months
  The within patient mean change from baseline to 6 months in Neck Disability Index scores. Scale of 0-50; 0-4 points (no disability), 5-14 points (mild disability), 15-24 points (moderate disability), 25-34 points (severe disability), 35-50 points (complete disability).
Neck Disability Index score change from baseline | Change from baseline to 12 months
  The within patient mean change from baseline to 12 months in Neck Disability Index scores.scores. Scale of 0-50; 0-4 points (no disability), 5-14 points (mild disability), 15-24 points (moderate disability), 25-34 points (severe disability), 35-50 points (complete disability).
Short Form Health Survey score change from baseline | Change from baseline to 6 months
  The within patient mean change from baseline to 6 months in Short Form Health Survey. Two summary scores are derived; the Physical component scale and the Mental component scale, each on a scale of 0-100, where the higher the score, the better the health.
Short Form Health Survey score change from baseline | Change from baseline to 12 months
  The within patient mean change from baseline to 12 months in Short Form Health Survey. The within patient mean change from baseline to 6 months in Short Form Health Survey. Two summary scores are derived; the Physical component scale and the Mental component scale, each on a scale of 0-100, where the higher the score, the better the health.
Numeric Pain scale change from baseline | Change from baseline to 6 months
  The within patient mean change from baseline to 6 months in Numeric Pain scale, where 0=no pain and 10=worst possible pain.
Numeric Pain scale change from baseline | Change from baseline to 12 months
  The within patient mean change from baseline to 12 months in Numeric Pain scale, where 0=no pain and 10=worst possible pain.
Single Assessment Numeric Evaluation improvement rating-modified | Mean at 6 months
  Mean improvement scores at 6 months, where -100=100% worse from baseline and 100=100% better or improved from baseline.
Single Assessment Numeric Evaluation improvement rating-modified | Mean at 12 months
  Mean improvement scores at 12 months, where -100=100% worse from baseline and 100=100% better or improved from baseline.
Adverse events | Thru 12 months post-procedure
  Any complication or adverse event
C1-C2 overhang | At least 6 months post-procedure
  Post-op DMX studies to quantify any reduction in C1-C2 overhang or ADI.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Centeno-Schultz Clinic
Locations (1):
- Centeno-Schultz Clinic, Broomfield, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centeno CJ, Elliott J, Elkins WL, Freeman M. Fluoroscopically guided cervical prolotherapy for instability with blinded pre and post radiographic reading. Pain Physician. 2005 Jan;8(1):67-72. PMID 16850045
- [Background] Panjabi MM, Crisco JJ 3rd, Lydon C, Dvorak J. The mechanical properties of human alar and transverse ligaments at slow and fast extension rates. Clin Biomech (Bristol). 1998 Mar;13(2):112-120. doi: 10.1016/s0268-0033(97)00053-3. PMID 11415778
- [Background] Rajwanshi A, Rohilla M, Singh P. Trans-oral fine needle aspiration cytology in cervical (C1 and C2) vertebral lesions: a novel diagnostic approach. Cytopathology. 2017 Feb;28(1):31-34. doi: 10.1111/cyt.12361. Epub 2016 Aug 3. PMID 27489015
- [Background] Centeno CJ, Pitts J, Al-Sayegh H, Freeman MD. Anterior cruciate ligament tears treated with percutaneous injection of autologous bone marrow nucleated cells: a case series. J Pain Res. 2015 Jul 31;8:437-47. doi: 10.2147/JPR.S86244. eCollection 2015. PMID 26261424